CLINICAL TRIAL: NCT07123714
Title: Effect of Preoperative Nebulized Magnesium Sulfate on Post-intubation Stress Response in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effect of Nebulized Magnesium Sulfate on Post-intubation Stress Response in Patients Undergoing Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17101959
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Sore Throat
Keywords: Magnesium sulfate nebulization; postoperative sore throat; Post-intubation sore throat; Post-intubation stress response
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized magnesium sulfate group (Experimental): Patients will receive nebulized magnesium sulfate in 5 ml (250 mg) over 15 min.
  Interventions: Procedure: Nebulization of magnesium sulfate
- control group (No Intervention): Patients will receive nebulized normal saline 5ml, 15 minutes preoperatively

INTERVENTIONS:
Procedure: Nebulization of magnesium sulfate — patient will be nebulized with 5 mg magnesium sulfate (5 ml) 15 minutes before induction of anesthesia
  Arms: Nebulized magnesium sulfate group

SUMMARY:
This randomized controlled double blinded study will be carried out on 140 patients underwent elective fit laparoscopic cholecystectomy at El-Rajhi Assiut University Hospital.

Inclusion criteria:

* 20-50 years old.
* Both sexes.
* American society of anesthesiologists (ASA) physical status I-II.
* Elective fit laparoscopic cholecystectomy

Exclusion criteria:

* Patient refusal.
* Patients with history of hypersensitivity to magnesium sulfate.
* Patients with coronary ischemic disease, atrioventricular block of any degree, known cardiac arrhythmias, heart failure on beta blockers or calcium channel blockers expected difficult intubation (Mallampati 4).
* Body mass index (BMI) > 40 kg/m2.

An online randomization program (http://www.randomizer.org) will be used to generate a random list and each patients' code will be kept in an opaque sealed envelope. Patients will be randomly allocated with 1:1 allocation ratio into two equal groups in a parallel manner:

* Group A: (N=70) Patients will receive nebulized magnesium sulfate in 5 ml (250 mg) over 15 min.
* Group B: (N=70) Patients received nebulized normal saline in 5 ml over 15 min, ending 5 min before the induction of anesthesia.

A. Preoperative assessment:

All patients will be subjected to the followings:

1. Demographic data collection (age, weight, height, BMI, and ASA).
2. Complete clinical examination.
3. Routine Laboratory investigations:

   * Random blood sugar.
   * Blood sample withdrawal for cortisol level at baseline 2ml intravenously. The sample will be sent to be centrifugated within 30 minutes and the serum will be separated and stored in -20°C till time of cortisol level by ELIZA technique.

DETAILED DESCRIPTION:
B. Intraoperatively:

SBP, DBP, HR, and blood glucose level will be measured at the following intervals: Baseline (before induction), after premedication (sedation), after induction, after ETT intubation, 3 min later, 6 min later.

Full monitoring data (Blood pressure every 3 minutes, ECG, Nanogram, and pulse oximeter) will be collected till 6 minutes then every 5 minutes. Random blood sugar will be tested 5 minutes pre-intubation, 3minutes and 5 minutes after intubation and recorded.

After end of nebulization, sedation with 2 mg midazolam and IV fluids (10 ml/kg) were infused to avoid tachycardia of dehydration and fear of surgery. Then, we proceed on general anesthesia through Propofol titration + fentanyl 100 mcg + Cis-atracurium 0.15 mg/kg. Endotracheal intubation with cuffed tube and mechanical ventilation with mild increase in respiratory rate 14-16/min to overcome CO2 peritoneal insufflation.

All patients will receive intraoperatively, nalbuphine 0.1 mg/kg + ketorolac 60 mg + paracetamol IV 1 g. Dexamethasone 4mg + Ondansetron 4mg will receive to all patients for prophylaxis against postoperative nausea and vomiting.

After 10 minutes of intubation, a second 2ml IV blood sample will be withdrawn for cortisol level. The centrifugation, serum separation, storage and ELIZA analysis will be done as the baseline sample described above.

C. Postoperative:

After end of surgery, cessation of inhalational anesthesia and reversal of muscle relaxation with neostigmine 2.5 mg+ Atropine 1mg is done. Consumption of isoflurane intraoperatively is recorded. Post operative assessment for pain using Visual Analogue Scale (VAS) will be assessed 2 hours after recovery. VAS is presented as a website10 cm straight line ruler reflecting the extremes of "no pain" equals 0 and "worst pain at the other end(at 10cm), while in between the intensity of pain is represented by corresponding facies.

Time for recovery after stop of isoflurane is estimated. Hypertension is considered when the BP values are 20% above baseline values or SBP > 140 mmHg. Hypotension is considered when BP values are lower than 20% of baseline or SBP < 90 mmHg and will be treated with 10-20 mg ephedrine. Tachycardia will be considered when HR is higher than 20% of baseline or HR > 100 bpm. Bradycardia is considered when HR values are lower than 50 bpm, treated by I.V. atropine 0.02 mg/kg respiratory depression (the SpO2 < 95% and need O2 supplementation), and postoperative nausea and vomiting (PONV) is treated by ondansetron 0.1 mg/kg IV.

Measurements:

* Demographic data.
* Hemodynamics variables like SBP, DBP, HR, and blood glucose level are measured at the following intervals: Baseline (before induction), after premedication (sedation), after induction, after ETT intubation, 3 min later, 6 min later.
* Visual Analog Scale (VAS) is assessed.
* Side effects are recorded

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) physical status I-II.
* Elective fit laparoscopic cholecystectomy

Exclusion Criteria:

* • Patient refusal.

  * Patients with history of hypersensitivity to magnesium sulphate.
  * Patients with coronary ischemic disease, atrioventricular block of any degree, known cardiac arrhythmias, heart failure on beta blockers or calcium channel blockers expected difficult intubation (Mallampati 4).
  * Body mass index (BMI) > 40 kg/m2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Difference between preoperative cortisol level and 6minutes after intubation | 6 minutes after intubation
  cortisol level will be measured preoperatively and 6 minutes after intubation then calculation of the difference between them then comparison between both groups

SECONDARY OUTCOMES:
NRS for sore throat postoperatively | 24 hours
  Pain will be assessed by numeric rating scale NRS asking the patient about his degree of pain graded from 0 to 10 in which 0 refers to no pain at all and 10 refers to the worst pain experienced in life
4 grade scale | 24 hours postoperatively
  examination of the degree of laryngeal dysfunction due to sore throat into 4 grades: grade 1 refers to no pain, 2 refers to pain during swallowing, 3 =continuous pain and increases with swallowing and 4 refers to severe pain that hinders eating and necessitates urgent treatment.
Random blood sugar RBS | 6 minutes after intubation
  RBS refers to stress and known to increase with stress

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yadav M, Chalumuru N, Gopinath R. Effect of magnesium sulfate nebulization on the incidence of postoperative sore throat. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):168-71. doi: 10.4103/0970-9185.173367. PMID 27275043
- [Background] 2. Gutiérrez-Román, C.I., O. Carrillo-Torres and E.S. Pérez-Meléndez, Uses of magnesium sulfate in anesthesiology. Revista médica del Hospital General de México, 2022. 85(1): p. 25-33, .
- [Background] Chen Z, Zuo Z, Zhang L, Gong M, Ye Y, Jin Y, Zhao X. Postoperative Sore Throat After Tracheal Intubation: An Updated Narrative Review and Call for Action. J Pain Res. 2025 May 6;18:2285-2306. doi: 10.2147/JPR.S498933. eCollection 2025. PMID 40352818